CLINICAL TRIAL: NCT04070482
Title: The Impact of in Utero and Breastfeeding Exposure to Tenofovir on Renal Function in HIV-exposed Uninfected Children in Cameroon: The PREVENT-IT Study
Brief Title: Impact of in Utero and Breastfeeding Exposure to Tenofovir on Renal Function in HIV-exposed Uninfected Children
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Yaounde 1 (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Principal Investigator, Gabriel Loni Ekali, Research Fellow, University of Yaounde 1
Other Study IDs: 2016/449-LON
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Renal Injury
Keywords: Tenofovir; HIV-exposed infants; renal injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Mothers: Peripheral blood (delivery) Infants: Coord blood, urine, peripheral blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HIV-exposed uninfected infants: These are children to women who are living with HIV but who are not infected with the virus (HIV PCR results at 6 weeks is negative)
  Interventions: Other: Tenofovir exposure in utero and during breastfeeding
- HIV-unexposed uninfected infants: These are children born to women who are not infected with HIV

INTERVENTIONS:
Other: Tenofovir exposure in utero and during breastfeeding — Exposed in utero and during breastfeeding to Tenofovir-containing antiretroviral drugs
  Groups: HIV-exposed uninfected infants

SUMMARY:
The goal of this project is to determine whether and how in utero exposure to Tenofovir affects renal function in HIV-exposed uninfected infants

DETAILED DESCRIPTION:
There is a growing use of Tenofovir (TDF) in sub-Saharan Africa with the use of Option B+ for prevention of mother-to-child HIV transmission. TDF has been associated to renal function abnormalities both in macaques and HIV-infected adults and infants. Therefore concerns have been raised about its renal safety in exposed infants of women on Option B+. Data for HEU is sparse and routine measures of renal function (creatinine, proteinuria), may not be appropriate to detect TDF-associated renal injury early. The goal of our study is to assess whether TDF use in pregnancy and breastfeeding affects the function of the kidney function of the child. Pregnant women who consent during their first antenatal consultation to take antiretroviral drugs for PMTCT after testing positive, will be enrolled and followed till birth, for adherence using HPLC. Their terms infants who are HIV negative by DNA PCR at 6 weeks (HEU), will have urine collected at 1.5, 3, 6, 9 months. Using appropriate and more sensitive markers (RBP4, KIM1, NAG, β2M), proximal tubular function will be assessed in 159 HEU infants and same number of controls. Nutritional status and drug history data will be collected for both mother and child. RBP, KIM1, β2M will be measured using XMAP assay while ELISA will be used for NAG according to manufacturer recommendations. Creatinine, phosphates and urinary tract infection will be measured using standard methods. Values of these markers will be compared between the 2 groups. Results will confirm/infirm renal safety of TDF in pregnancy, improve prevention of long term renal injury through early detection, contribute to promote development of routine rapid diagnostic tests for acute renal tubular injury

ELIGIBILITY:
Inclusion Criteria:

* Mothers

  1. HIV seropositive pregnant women on Option B+ protocol containing TDF.
  2. HIV seronegative pregnant women
  3. Pregnant women who provide informed consent.
  4. Woman is living in Yaounde and is not planning to relocate in the next 2 years. Children

  <!-- -->

  1. Children born to HIV-infected mothers (and HIV-uninfected mothers for controls).
  2. TDF- and HIV-exposed in utero (and age-matched unexposed controls).
  3. HIV negative after birth by DNA PCR 4.0 to 12 months of age (included in study at birth and followed up till 12 months)

Exclusion Criteria:

* Refusal of parent(s) to give consent

Max Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Our study population will be primarily made up of mother-infant pairs with and without infant exposure in utero to TDF and HIV
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Difference in urinary RBP, NAG, KIM-1and B2M levels at birth between neonates born to mothers living with HIV, exposed in utero to TDF and those born to mothers without HIV and not exposed to TDF | Birth
  In urine samples collected at birth from HIV-EU TDF-exposed neonates and an equal number of TDF-unexposed controls, RBP, KIM-1, B2M will be measured using multianalyte platform (xMAP) assay, while NAG will be measured using ELISA. Levels of these correlates of proximal tubular function will be compared between the two groups, adjusting for confounders
Difference in urinary RBP, NAG, KIM-1and B2M levels after birth and within the first year of life between HEU infants, exposed in utero to TDF and HUU infants, not exposed to TDF | 0 to 12 months
  Trends in urinary RBP:Cr, NAG:Cr, KIM-1 and B2M will be tracked during and beyond breastfeeding between HIV-EU TDF+ and unexposed controls by conducting serial measurements of these markers at 6 weeks then 3, 6, 12 months using same methods described in outcome 1

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel L Ekali, MD,MH, Principal Investigator — University of Yaounde 1
Locations (3):
- Cameroon (3):
  - CASS, Yaoundé
  - Cité Verte DH, Yaoundé
  - Efoulan DH, Yaoundé